CLINICAL TRIAL: NCT03854292
Title: ICSI Pregnancy Outcomes Following Hysteroscopic Tubal Electrocoagulation Versus Laparoscopic Tubal Disconnection for Patients With Hydrosalpinges
Brief Title: Hydrosalpinx Management Before Intracytoplasmic Sperm Injection
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Abdalla, Principal Investigator, Cairo University
Other Study IDs: tubal disconnection
Record Dates: First submitted 2019-02-23; First posted 2019-02-26 (Actual); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Hydrosalpinx

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hysteroscopic tubal electrocoagulation: Unilateral or bilateral electrocoagulation of the cornual end of the tube and the surrounding part of the uterine horn was performed using a hysteroscopic electrocoagulating roller ball
  Interventions: Procedure: Hysteroscopic tubal electrocoagulation
- Laparoscopic tubal disconnection: Coagulation of the mid isthmus region of the affected Fallopian tube, with the bipolar forceps. using direct current that was no greater than 25 Watts.
  Interventions: Procedure: Hysteroscopic tubal electrocoagulation

INTERVENTIONS:
Procedure: Hysteroscopic tubal electrocoagulation — Unilateral or bilateral electrocoagulation of the cornual end of the tube and the surrounding part of the uterine horn was performed using a hysteroscopicelectrocoagulating roller ball.

SUMMARY:
ICSI pregnancy outcomes following hysteroscopic tubal electrocoagulation versus laparoscopic tubal disconnection for patients with hydrosalpinges

DETAILED DESCRIPTION:
Tubal factor of infertility resulting from various forms of tuboperitoneal damage remains an extremely common cause of female infertility, accounting for more than 35% of all cases of female infertility. Probably the most severe form of tubal pathology is hydrosalpinx. Hydrosalpinx is a Greek word that means a Fallopian tube filled with water or fluid. Patients with hydrosalpinges have been identified as a subgroup with significantly lower implantation and pregnancy rates than patients with other tubal pathologies. An increased risk for early pregnancy loss and increased risk for ectopic pregnancies was reported, and many studies confirmed that the presence of hydrosalpinx significantly impairs in vitro fertilization (IVF) outcome as well.

Patients with a hydrosalpinx have been found to have significantly poorer outcomes of IVF than do patients with tubal factor infertility but no hydrosalpinx .

Hydrosalpinges in infertile women reduce the success of IVF by 50 % .

The harmful effect of a hydrosalpinx on pregnancy rates after IVF has been attributed to mechanical washout of the transferred embryos by tubal-uterine reflux of the hydrosalpinx fluid .

Additionally, a hydrosalpinx might disturb endometrial receptivity: integrins, the best endometrial markers, show decreased expression in cases of hydrosalpinx .

Altered endometrial blood flow has also been proposed as a possible factor causing decreased rates of implantation.

Any surgical interventions that disrupt tubal-uterine communication in affected tubes might improve pregnancy rates .

Laparoscopic salpingectomy was the most popular treatment option offered by the clinicians, followed by open salpingectomy, salpingostomy, proximal tubal occlusion and transvaginal ultrasonographic guided hydrosalpinx aspiration either before or during oocyte retrieval.The latest treatment option introduced was proximal occlusion of the hydrosalpinx by hysteroscopic placement of microinserts. Clinicians would still perform open salpingectomy. The possible explanation for this could be the lack of training in endoscopic surgery and/or that patients with tubal disease may have significant pelvic adhesions necessitating open surgery.

Laparoscopic salpingectomy or tubal ligation has been shown to improve IVF outcomes for patients with a hydrosalpinx.

However, this procedure has many drawbacks, including its invasiveness, the possibility of surgical injury (e.g. visceral injury, vascular damage, or unintended laparotomy), the potential risks from general anesthesia, and technical difficulty if there are pelvic adhesions .

The proximal occlusion of a hydrosalpinx by hysteroscopy might offer a feasible therapeutic alternative when laparoscopy is technically difficult or contraindicated,with the advantage of hysteroscopic procedures of faster recovery, less hospitalization and rapid return to work, and in the future it might be done in the outpatient clinic as an office procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age from 20 to 35 years
* Primary or secondary infertility.
* Diagnosis of hydrosalpinx; diagnosed by HSG and TV U/S.
* Necessity of an IVF procedure.

Exclusion Criteria:

* Patients with uterine factor infertility.
* Medical or surgical conditions contraindicating pregnancy.
* Poor responders according to reference criteria.
* Cases of polycystic ovary disease.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 50 patients who have unilateral or bilateral hydrosalpinges identified on hysterosalpingography and vaginal ultrasonography, and who are undergoing IVF.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
proximal tubal occlusion Success rate . | 15 months
  proximal tubal occlusion Success rate among two groups detected by Hysterosalpingogram.

SECONDARY OUTCOMES:
Pregnancy rate among the two groups. | 15 months
  Chemical Pregnancy rate among the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Strandell A, Waldenstrom U, Nilsson L, Hamberger L. Hydrosalpinx reduces in-vitro fertilization/embryo transfer pregnancy rates. Hum Reprod. 1994 May;9(5):861-3. doi: 10.1093/oxfordjournals.humrep.a138606. PMID 7929732
- [Background] Strandell A, Lindhard A, Waldenstrom U, Thorburn J, Janson PO, Hamberger L. Hydrosalpinx and IVF outcome: a prospective, randomized multicentre trial in Scandinavia on salpingectomy prior to IVF. Hum Reprod. 1999 Nov;14(11):2762-9. doi: 10.1093/humrep/14.11.2762. PMID 10548619
- [Background] Puttemans P, Campo R, Gordts S, Brosens I. Hydrosalpinx and ART: hydrosalpinx--functional surgery or salpingectomy? Hum Reprod. 2000 Jul;15(7):1427-30. doi: 10.1093/humrep/15.7.1427. PMID 10875845
- [Background] Mijatovic V, Veersema S, Emanuel MH, Schats R, Hompes PG. Essure hysteroscopic tubal occlusion device for the treatment of hydrosalpinx prior to in vitro fertilization-embryo transfer in patients with a contraindication for laparoscopy. Fertil Steril. 2010 Mar 1;93(4):1338-42. doi: 10.1016/j.fertnstert.2008.11.022. Epub 2009 Jan 14. PMID 19147140
- [Background] Savaris RF, Pedrini JL, Flores R, Fabris G, Zettler CG. Expression of alpha 1 and beta 3 integrins subunits in the endometrium of patients with tubal phimosis or hydrosalpinx. Fertil Steril. 2006 Jan;85(1):188-92. doi: 10.1016/j.fertnstert.2005.06.039. PMID 16412752
- [Background] Hammadieh N, Afnan M, Evans J, Sharif K, Amso N, Olufowobi O. A postal survey of hydrosalpinx management prior to IVF in the United Kingdom. Hum Reprod. 2004 Apr;19(4):1009-12. doi: 10.1093/humrep/deh133. Epub 2004 Mar 11. PMID 15016787
- [Background] Kontoravdis A, Makrakis E, Pantos K, Botsis D, Deligeoroglou E, Creatsas G. Proximal tubal occlusion and salpingectomy result in similar improvement in in vitro fertilization outcome in patients with hydrosalpinx. Fertil Steril. 2006 Dec;86(6):1642-9. doi: 10.1016/j.fertnstert.2006.05.032. Epub 2006 Oct 25. PMID 17069813
- [Background] El-Mazny A, Abou-Salem N, Hammam M, Saber W. Hysteroscopic tubal electrocoagulation versus laparoscopic tubal ligation for patients with hydrosalpinges undergoing in vitro fertilization. Int J Gynaecol Obstet. 2015 Sep;130(3):250-2. doi: 10.1016/j.ijgo.2015.04.039. Epub 2015 Jul 2. PMID 26140948
- [Background] Parihar M, Mirge A, Hasabe R. Hydrosalpinx functional surgery or salpingectomy? The importance of hydrosalpinx fluid in assisted reproductive technologies. J Gynecol Endosc Surg. 2009 Jan;1(1):12-6. doi: 10.4103/0974-1216.51903. PMID 22442504
- [Background] Stadtmauer LA, Riehl RM, Toma SK, Talbert LM. Cauterization of hydrosalpinges before in vitro fertilization is an effective surgical treatment associated with improved pregnancy rates. Am J Obstet Gynecol. 2000 Aug;183(2):367-71. doi: 10.1067/mob.2000.107671. PMID 10942471